CLINICAL TRIAL: NCT05160012
Title: Peer Comparison Feedback to Providers to Improve Hypertension Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 849584
Record Dates: First submitted 2021-11-09; First posted 2021-12-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will not receive peer comparison messages and will continue with usual care.
- Intervention (Experimental): This group will receive peer comparison messages.
  Interventions: Behavioral: Peer Comparison Message

INTERVENTIONS:
Behavioral: Peer Comparison Message — In addition to usual care, PCPs will receive a monthly report as an EPIC in basket message describing what category they are in:
  1. If HTN control rate <50th percentile, PCP is told they are below median
  2. If HTN control rate is between 50-89th percentile , PCP is told they are below top performer
  3. If HTN control rate is between 90-100th percentile, PCP is told they are a high performer
  Arms: Intervention

SUMMARY:
As part of a roll out of new payment model for physicians based on hypertension control, the investigators will evaluate a monthly peer comparison message to Primary Care Providers at Penn Medicine Lancaster to see whether provider engagement with patients' overall hypertension management increases, as measured by new or increasing doses of anti-hypertensive medications.

DETAILED DESCRIPTION:
Hypertension (HTN) affects about 30% of US adults, and effective treatment that reduces long-term risk of subsequent cardiovascular disease is widely available; however, only about half of adults maintain good control. HTN control requires diagnosis, initiation of treatment, adherence to medications, and titration of medications. The investigators' prior work from Way2Text and SupportBP showed that there is significant clinical inertia in escalating medications for HTN through increasing dosage or adding new medications.

Prior studies have shown that providing feedback to providers with peer comparison data can leverage social norms to improve evidence-based practices in antibiotic and statin prescribing. Penn Medicine Lancaster General Primary Care is rolling out a Hypertension Control Implementation Plan (HCIP) as an initiative to improve hypertension control through creation of a clinic-based pathway to identify patients with hypertension, appropriately measure blood pressure, and prescribe medications to reduce blood pressure. Busy PCPs have competing demands of care, so there is an opportunity to leverage peer comparison to nudge providers to adhere to the HCIP and intensify medications.

The study design is a stratified parallel-group cluster-randomized trial. PCPs will be randomized in a 1:1 ratio, stratified by practice, to either: 1) Control: Usual Care- This will include the standard HCIP roll-out, and PCPs can access their HTN control rates using the existing EPIC dashboard.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Providers who have at =>30 patients hypertension as determined by the HTN quality metric
* Patients aged 18-85 with hypertension in their encounter diagnosis within the last 2 years (office visits, ED/Urgent Care, Hospital, Hospital Encounter, and Prenatal Visit)
* Patients will be counted in the denominator of the quality metric if they have both systolic and diastolic BP measures from an encounter with their PCP department within the last year (including office visits, well child, prenatal visit, consult visit, confidential, e-visit, nursing only, home/offsite visit, and telemedicine) that is >140 for systolic BP and >90 diastolic BP

Exclusion Criteria:

* Primary Care Providers includes providers with <30 patients in the HTN quality metric
* Patients will be excluded if they are 66 and older with a frailty diagnosis and those with an advanced illness diagnosis within the past year; 81 and older with frailty diagnosis within the past year
* It also excludes patients with end stage renal disease (indicated by evaluation of the GFR, diagnosis of end stage renal disease in last year, dialysis received in last year, or renal transplant) and patients with a pregnancy diagnosis in the last 9 months
* It also excludes patients with an end of life indicator (comfort care encounter in last year, comfort care noted in problem list in last year, and comfort care/palliative care procedures in last year)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in new hypertensive medication prescriptions or an increased dose of hypertensive medication | 6 months
  Change in new hypertensive medication prescriptions or an increased dose of hypertensive medication from baseline to the follow up period, as measured by the proportion of patients with a new prescription or dose placed for hypertensive medications in the electronic health record (EHR) from baseline to follow-up

SECONDARY OUTCOMES:
Change in hypertension control percentage | 6 months
  Change in hypertension control percentage from baseline to follow up period, as measured by percentage increases in a hypertension quality improvement report that is provided to physicians in the electronic health record (EHR) and reflects rate of hypertension control across all patients under the care of that physician.

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD,MBA,MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States